CLINICAL TRIAL: NCT00428038
Title: Assessment of the Pulmonary Diffusion Capacity in Healthy Infants and Infants With Chronic Lung Disease
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: 0309-15
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Infant, Premature; Bronchopulmonary Dysplasia; Asthma
Keywords: Infant, Premature; Bronchopulmonary Dysplasia; Asthma
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Group 1:
  Infants born prematurely at a gestational age < 32 weeks with a diagnosis of chronic lung disease. Subjects will be evaluated at a corrected-age between 1 month and 24 months when they are clinically stable and free of acute respiratory symptoms for > 3 weeks. Subjects will be excluded for the following reasons:
  1. Oxygen requirements
  2. Congenital heart disease
- 2: Group 2:
  Infants born prematurely at a gestational age < 32 weeks without a diagnosis of chronic lung disease. Subjects will be evaluated at a corrected-age between 1 month and 24 months when they are clinically stable and free of acute respiratory symptoms for > 3 weeks. Subjects will be excluded for the following reasons:
  1. Oxygen requirements
  2. Congenital heart disease
- 3: Group 3:
  Infants born full term at a gestational age > 37 weeks. Subjects will be evaluated at a corrected-age between 1 month and 24 months when they are clinically stable and free of acute respiratory symptoms for > 3 weeks. Subjects will be excluded for the following reasons:
  1. Hospitalization for a respiratory illness
  2. History of wheezing, asthma, or treatment with asthma medications
  3. Congenital heart disease

SUMMARY:
The purpose of this study is to evaluate how easily gas can be taken up by the lung. We are comparing infants born premature <32 weeks gestation to infants born full term >37 weeks. We hope to evaluate the differences between the two groups in order to learn more about premature lung growth and development.

DETAILED DESCRIPTION:
We hypothesize that infants who were born prematurely but are clinically without chronic respiratory disease have a lower lung diffusion capacity than healthy infants born at full term, when evaluated at comparable post-conception ages. In addition, prematurely born infants that develop chronic lung disease have an even lower diffusion capacity than healthy premature infants and full term infants. A lower diffusion capacity, when normalized to lung volume, would be consistent with decreased alveolarization and alveolar surface area in the infants born prematurely. We will study the age range of 1 to 24 month as this represents the period of rapid lung growth.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 Infants born at < 32 weeks gestation with Chronic lung disease
* Group 2 Infants born at <32 weeks gestation without Chronic lung disease
* Group 3 Infants born full term at >37 weeks

Exclusion Criteria:

* Group 1 and Group 2--No heart disease, no oxygen requirement
* Group 3--No hospitalization for respiratory illness, No asthma, No heart disease, No history of wheezing, asthma or treatment with asthma medications.

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Recruitment for premature infants were through Infant Lung Disease clinic at Riley Hospital for Children and IU NICU. Healthy full term infants were recruited through advertisements in local newspapers.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2004-02; Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Tepper, MD, PhD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States